CLINICAL TRIAL: NCT03512509
Title: Comparison of Low GI and High GI Potatoes in Relation to Satiety - a Randomised Control Trial
Brief Title: Comparison of Low GI and High GI Potatoes in Relation to Satiety (POSAT)
Acronym: POSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Birgitte Raben (Other)
Responsible Party: Sponsor-Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B344
Record Dates: First submitted 2018-03-15; First posted 2018-04-30 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Single-blind randomized crossover
Who Masked: Participant
Masking Description: Subjets will not be aware of which test meal they will recieve first, and are not able to distinguish between the two potatoes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Low glycaemic potato
  Interventions: Other: Low glycaemic potato
- B (Experimental): High glycaemic potato
  Interventions: Other: High glycaemic potato

INTERVENTIONS:
Other: Low glycaemic potato — The Carisma potato variety is used as the low glycaemic index potato.
  Arms: A
Other: High glycaemic potato — The Arizona potato variety is used as the high glycaemic index potato.
  Arms: B

SUMMARY:
The study is a single-blind, randomised crossover study, investigating how a high glycaemic potato affects satiety in humans compared to a low glycaemic potato. This is done to shed further light on the discussion about whether potatoes with a high glycaemic index increases the risk of overweight and obesity and thus indirectly type 2 diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
The POSAT study follows a single-blinded randomized crossover design. Each subject will have two separate intervention days with at least a six-day washout period in between. On the two intervention days the subjects will be randomized into receiving a breakfast containing isocaloric amounts of either low or high GI potatoes. VAS will be measured 5 minutes before the meal, immediately after the meal is consumed and in intervals of 30 minutes thereafter until 2,5 hours after the initial meal. After this the subjects will be served a standardized homogenous ad libitum meal. The amount of food consumed will be registered. The subjects will be asked to fast for 8-10 hours prior to the trial days and abstain from vigorous physical activity and alcohol consumption for 2 days prior to each trial day. The trial will be conducted over a total of 8 days with 5-6 study subjects pr. trial day. The trial days will be spread out over a total of 2 weeks to allow for a 1-week washout period between trial days for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Body mass index (BMI) 18-27 kg/m2
* Age 18-40 years
* Signed informed consent
* Able to eat 500 grams of potato for breakfast

Exclusion Criteria:

* Chronic diseases as diabetes, cardiovascular diseases or other chronic metabolic diseases, which could affect the results.
* Use of daily prescription medicine (mild analgesics and antihistamines are allowed).
* Use of medicine or dietary supplements that can affect ones appetite one month before the start of the study.
* Smoking or have been smoking or using any nicotine products (gum or e-cigarette) within the last 3 months. Irregular smoking is allowed.
* Elite athletes defined as doing >10 hours of strenuous physical activity per week.
* Participation in other clinical studies <1 month before or during the study.
* Inability, physically or psychologically, to comply with the procedures required by the study protocol. Judged by the investigators.
* Any food allergies.
* Weight change of ±3 kg from screening to the trial has been conducted.
* Inability to complete the trial within 3 months after screening.
* Unable to fast 8-10 hours before the trial days.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Subjective satiety evaluation | 3 hours
  Visual Analogue Scale (100mm) filled out by subjects to describe satiety.

SECONDARY OUTCOMES:
Hunger, fullness, and prospective food consumption | 3 hours
  Visual Analogue Scale (100mm) filled out by subjects to describe hunger, fullness, and prospective food consumption.
Energy consumed in Ad libitum meal | 30 minutes
  Energy intake (kJ) meassured by weighing of food consumed during a ad libitum meal.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Raben, Professor, Principal Investigator — Department of Nutrition, Sports and Exercise, University of Copenhagen
Locations (1):
- University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided